CLINICAL TRIAL: NCT01001104
Title: Assessment of Dose-Dependent Effects of LY2189265 on Glycemic Control in Japanese Patients With Type 2 Diabetes
Brief Title: A Study of LY2189265 in Japanese Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12840; H9X-JE-GBCZ (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-10-22; First posted 2009-10-23 (Estimated); Results first posted 2015-09-28 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Metabolic Diseases; Glucose Metabolism Disorders; Diabetes; GLP-1; Lilly
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Metabolic Diseases; Glucose Metabolism Disorders; Diabetes Mellitus | interventions — dulaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 0.75 mg LY2189265 (Experimental)
  Interventions: Drug: LY2189265
- 0.5 mg LY2189265 (Experimental)
  Interventions: Drug: LY2189265
- 0.25 mg LY2189265 (Experimental)
  Interventions: Drug: LY2189265
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY2189265 — Administered by subcutaneous (SC) injection, once weekly (QW) for 12 weeks.
  Arms: 0.25 mg LY2189265; 0.5 mg LY2189265; 0.75 mg LY2189265
Drug: Placebo — Administered by SC injection, QW for 12 weeks.
  Arms: Placebo

SUMMARY:
The main purpose of this study is to assess dose-response characteristics in Japanese patients with Type 2 Diabetes taking LY2189265 monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Japanese patients with type 2 diabetes with a body mass index (BMI)≥18.5 kilograms per square meter (kg/m^2) but <40.0 kg/m^2.
* Patients who are oral antidiabetic drug (OAD) naïve or are taking OAD monotherapy except for a dipeptidyl peptidase-4 inhibitor (DPP-IV) and are willing to discontinue their OAD.
* Patients who are OAD naïve with screening glycosylated hemoglobin (HbA1c) value of 7.0% to 9.5% and randomization HbA1c value of 7.0% to 9.5%, or who are taking OAD monotherapy with screening HbA1c value of 6.0% to 8.5% and randomization HbA1c value of 7.0% to 9.5%.
* Patients who have, in the opinion of the investigator, a stable weight during the 12 weeks prior to screening.

Exclusion Criteria:

* Patients who are currently taking prescription medications to promote weight loss
* Patients who are receiving chronic systemic glucocorticoid therapy, or have received such therapy within 4 weeks immediately prior to screening.
* Patients who have a known clinically significant gastrointestinal disorder, have undergone excision of all or any part of the gastrointestinal tract, have undergone gastric bypass surgery for treatment of obesity, or chronically take drugs that directly influence gastrointestinal motility.
* Patients who have poorly controlled hypertension, renal artery stenosis, or evidence of labile blood pressure including symptomatic postural hypotension.
* Patients who have obvious clinical signs or symptoms of pancreatitis, a history of chronic pancreatitis or acute pancreatitis. Patients who have amylase and/or lipase of 1.5 times or more the upper limit of the reference range.
* Have a family history, obvious clinical signs, or symptoms of medullary carcinoma of thyroid.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2009-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9AM - 5PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (6):
- Japan (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kochi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo

RESULTS

PARTICIPANT FLOW:
Groups:
- 0.75 mg LY2189265: Administered by subcutaneous (SC) injection, once weekly (QW) for 12 weeks.
- 0.5 mg LY2189265; 0.25 mg LY2189265; Placebo: Administered by SC injection, QW for 12 weeks.
Period: Overall Study
Arm/Group | 0.75 mg LY2189265 | 0.5 mg LY2189265 | 0.25 mg LY2189265 | Placebo
Started | 35 | 37 | 36 | 37
Completed | 33 | 36 | 35 | 34
Not Completed | 2 | 1 | 1 | 3
Not completed — Adverse Event | 2 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Entry Criteria Not Met | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.75 mg LY2189265 | 0.5 mg LY2189265 | 0.25 mg LY2189265 | Placebo | Total
Number analyzed (Participants) | 35 | 37 | 36 | 37 | 145
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.23 (7.80) | 52.50 (9.17) | 52.26 (8.82) | 51.70 (9.67) | 52.17 (8.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 14 | 9 | 8 | 38
  Male | 28 | 23 | 27 | 29 | 107
Race/Ethnicity, Customized [Number; unit: participants]
  Japanese | 35 | 37 | 36 | 37 | 145
Region of Enrollment [Number; unit: participants]
  Japan | 35 | 37 | 36 | 37 | 145
Percentage of Glycosylated Hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin] | 8.01 (0.63) | 7.98 (0.66) | 8.05 (0.66) | 7.98 (0.64) | 8.00 (0.64)
Fasting Blood Glucose (FBG) [Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)] | 156.51 (26.43) | 150.95 (29.31) | 158.75 (35.62) | 159.65 (33.29) | 156.45 (31.26)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at 12 Weeks
Description: Change in HbA1c from baseline following 12 weeks of therapy (that is, HbA1c at week 12 minus HbA1c at baseline). Changes in HbA1c were analyzed by a mixed model repeated measures (MMRM) model that included dose, pre-study therapy, body mass index (BMI) group at baseline, baseline value, visit, and dose*visit, where the participant was treated as a random effect.
Time Frame: Baseline, 12 weeks
Population: Full analysis set: All randomized participants who received at least 1 dose of the study drug.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage glycosylated hemoglobin
Arm/Group | 0.75 mg LY2189265 | 0.5 mg LY2189265 | 0.25 mg LY2189265 | Placebo
Number analyzed (Participants) | 34 | 37 | 36 | 36
percentage glycosylated hemoglobin | -1.35 [-1.53 to -1.18] | -1.15 [-1.32 to -0.98] | -0.90 [-1.07 to -0.73] | -0.18 [-0.36 to -0.01]
Statistical Analysis 1: Comparison: 0.75 mg LY2189265 vs 0.5 mg LY2189265 vs 0.25 mg LY2189265 vs Placebo; Test type: Superiority or Other; p < .001, Mixed Models Analysis — This is the p-value for the linear trend test at 12 weeks
Statistical Analysis 2: Comparison: 0.25 mg LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Least Squares Mean Difference = -0.72
Statistical Analysis 3: Comparison: 0.5 mg LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Least Squares Mean Difference = -0.97
Statistical Analysis 4: Comparison: 0.75 mg LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Least Squares Mean Difference = -1.17

2. Secondary Outcome: Percentage of Participants Achieving Glycosylated Hemoglobin (HbA1c)<7% up to 12 Weeks
Description: Percentage of participants who achieved HbA1c<7% up to the 12-week endpoint.
Time Frame: up to 12 weeks
Population: All randomized participants who received at least 1 dose of the study drug, last observation carried forward (LOCF).
Measure: Number; unit: percentage of participants
Arm/Group | 0.75 mg LY2189265 | 0.5 mg LY2189265 | 0.25 mg LY2189265 | Placebo
Number analyzed (Participants) | 35 | 37 | 36 | 37
percentage of participants | 77.1 | 59.5 | 47.2 | 10.8
Statistical Analysis 1: Comparison: 0.75 mg LY2189265 vs 0.5 mg LY2189265 vs 0.25 mg LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Armitage — This is the p-value from the Cochran-Armitage trend test
Statistical Analysis 2: Comparison: 0.25 mg LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 3: Comparison: 0.5 mg LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 4: Comparison: 0.75 mg LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Fisher Exact

3. Secondary Outcome: Percentage of Participants Achieving Glycosylated Hemoglobin (HbA1c)<6.5% up to 12 Weeks
Description: Percentage of participants achieving HbA1c<6.5% up to the 12-week endpoint.
Time Frame: up to 12 weeks
Population: All randomized participants who received at least 1 dose of the study drug, last observation carried forward (LOCF).
Measure: Number; unit: percentage of participants
Arm/Group | 0.75 mg LY2189265 | 0.5 mg LY2189265 | 0.25 mg LY2189265 | Placebo
Number analyzed (Participants) | 35 | 37 | 36 | 37
percentage of participants | 34.3 | 24.3 | 8.3 | 2.7
Statistical Analysis 1: Comparison: 0.75 mg LY2189265 vs 0.5 mg LY2189265 vs 0.25 mg LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Armitage — This is the p-value from the Cochran-Armitage trend test
Statistical Analysis 2: Comparison: 0.25 mg LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.358, Fisher Exact
Statistical Analysis 3: Comparison: 0.5 mg LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.014, Fisher Exact
Statistical Analysis 4: Comparison: 0.75 mg LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Fisher Exact

4. Secondary Outcome: Change From Baseline in Fasting Blood Glucose (FBG) Values to 12 Weeks
Description: Change in FBG following 12 weeks of therapy (that is, FBG at week 12 minus FBG at baseline). The change in FBG was analyzed using a mixed model repeated measures (MMRM) model that included dose, pre-study therapy, body mass index (BMI) group at baseline, baseline value, visit, and dose*visit, where the participant was treated as a random effect.
Time Frame: Baseline, 12 weeks
Population: Full analysis set: All randomized participants who received at least 1 dose of the study drug.
Measure: Least Squares Mean (95% Confidence Interval); unit: milligrams per deciliter (mg/dL)
Arm/Group | 0.75 mg LY2189265 | 0.5 mg LY2189265 | 0.25 mg LY2189265 | Placebo
Number analyzed (Participants) | 35 | 37 | 36 | 37
milligrams per deciliter (mg/dL) | -37.48 [-47.00 to -27.97] | -28.55 [-37.68 to -19.41] | -29.21 [-38.45 to -19.97] | -9.00 [-18.39 to 0.38]
Statistical Analysis 1: Comparison: 0.75 mg LY2189265 vs 0.5 mg LY2189265 vs 0.25 mg LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — This is the p-value for the linear trend test at week 12
Statistical Analysis 2: Comparison: 0.25 mg LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis — Primary comparisons are based on the MMRM Least Squares (LS) Mean Value at week 12; Least Squares Mean Difference = -20.20
Statistical Analysis 3: Comparison: 0.5 mg LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis — Primary comparisons are based on the MMRM LS Mean Value at week 12; Least Squares Mean Difference = -19.54
Statistical Analysis 4: Comparison: 0.75 mg LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Primary comparisons are based on the MMRM LS Mean Value at week 12; Least Squares Mean Difference = -28.48

5. Secondary Outcome: Change From Baseline in the Mean Daily Blood Glucose (Based on Self-Monitoring Blood Glucose [SMBG]) at 12 Weeks
Description: SMBG levels were measured at the following 7 timepoints during the day: fasting prebreakfast, 2 hours postbreakfast, prior to lunch, 2 hours postlunch, prior to dinner, 2 hours postdinner, and prior to bed. The change in mean daily blood glucose was analyzed by a mixed model repeated measures (MMRM) model that included dose, pre-study therapy, body mass index (BMI) group at baseline, baseline value, and dose*visit, where the participant was treated as a random effect.
Time Frame: Baseline, 12 weeks
Population: Full analysis set: All randomized participants who received at least 1 dose of the study drug.
Measure: Least Squares Mean (95% Confidence Interval); unit: milligrams per deciliter (mg/dL)
Arm/Group | 0.75 mg LY2189265 | 0.5 mg LY2189265 | 0.25 mg LY2189265 | Placebo
Number analyzed (Participants) | 29 | 35 | 33 | 30
milligrams per deciliter (mg/dL) | -48.99 [-58.47 to -39.51] | -53.12 [-61.84 to -44.41] | -40.70 [-49.67 to -31.73] | -7.49 [-17.44 to 2.45]
Statistical Analysis 1: Comparison: 0.75 mg LY2189265 vs 0.5 mg LY2189265 vs 0.25 mg LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — This is the p-value for the linear trend test at week 12
Statistical Analysis 2: Comparison: 0.25 mg LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Primary comparisons are based on the MMRM Least Squares (LS) Mean Value at week 12; Least Squares Mean Difference = -33.20
Statistical Analysis 3: Comparison: 0.5 mg LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Primary comparisons are based on the MMRM LS Mean Value at week 12; Least Squares Mean Difference = -45.63
Statistical Analysis 4: Comparison: 0.75 mg LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Primary comparisons are based on the MMRM LS Mean Value at week 12; Least Squares Mean Difference = -41.49

6. Secondary Outcome: Change From Baseline in Total Body Weight at 12 Weeks
Description: Changes in body weight were analyzed by a mixed model repeated measures (MMRM) model that included dose, pre-study therapy, body mass index (BMI) group at baseline, baseline value, visit, and dose*visit, where the participant was treated as a random effect.
Time Frame: Baseline, 12 weeks
Population: Full analysis set: All randomized participants who received at least 1 dose of the study drug.
Measure: Least Squares Mean (95% Confidence Interval); unit: kilograms (kg)
Arm/Group | 0.75 mg LY2189265 | 0.5 mg LY2189265 | 0.25 mg LY2189265 | Placebo
Number analyzed (Participants) | 35 | 37 | 36 | 37
kilograms (kg) | -0.58 [-1.21 to 0.05] | -0.40 [-1.01 to 0.22] | 0.41 [-0.20 to 1.03] | -0.84 [-1.46 to -0.22]
Statistical Analysis 1: Comparison: 0.75 mg LY2189265 vs 0.5 mg LY2189265 vs 0.25 mg LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.987, Mixed Models Analysis — This is the p-value for the linear trend test at week 12
Statistical Analysis 2: Comparison: 0.25 mg LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis — Primary comparisons are based on the MMRM Least Squares (LS) Mean Value at week 12; Least Squares Mean Difference = 1.26
Statistical Analysis 3: Comparison: 0.5 mg LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.311, Mixed Models Analysis — Primary comparisons are based on the MMRM LS Mean Value at week 12; Least Squares Mean Difference = 0.45
Statistical Analysis 4: Comparison: 0.75 mg LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.556, Mixed Models Analysis — Primary comparisons are based on the MMRM LS Mean Value at week 12; Least Squares Mean Difference = 0.26

7. Secondary Outcome: Change From Baseline in Insulin Sensitivity Using the Updated Homeostasis Model Assessment Insulin Sensitivity (HOMA2-S) at 12 Weeks
Description: HOMA2-S is an estimated insulin sensitivity based on updated HOMA2 model. The HOMA2 model is a computer model that estimates insulin sensitivity (%S) as percentages of a normal reference population using simultaneously measured fasting plasma glucose and fasting insulin. Changes in HOMA2-S were analyzed by a mixed model repeated measures (MMRM) model that included dose, pre-study therapy, body mass index (BMI) group at baseline, baseline value, visit, and dose*visit, where the participant was treated as a random effect.
Time Frame: Baseline, 12 weeks
Population: Full analysis set: All randomized participants who received at least 1 dose of the study drug.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage insulin sensitivity (%S)
Arm/Group | 0.75 mg LY2189265 | 0.5 mg LY2189265 | 0.25 mg LY2189265 | Placebo
Number analyzed (Participants) | 32 | 32 | 33 | 33
percentage insulin sensitivity (%S) | -4.66 [-17.64 to 8.32] | -6.07 [-18.60 to 6.46] | 4.65 [-7.68 to 16.97] | 3.74 [-8.88 to 16.36]
Statistical Analysis 1: Comparison: 0.75 mg LY2189265 vs 0.5 mg LY2189265 vs 0.25 mg LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.202, Mixed Models Analysis — This is the p-value from the linear trend test at week 12
Statistical Analysis 2: Comparison: 0.25 mg LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.917, Mixed Models Analysis — Primary comparisons are based on the MMRM Least Squares (LS) Mean Value at week 12; Least Squares Mean Difference = 0.91
Statistical Analysis 3: Comparison: 0.5 mg LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.264, Mixed Models Analysis — Primary comparisons are based on the MMRM LS Mean Value at week 12; Least Squares Mean Difference = -9.81
Statistical Analysis 4: Comparison: 0.75 mg LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.346, Mixed Models Analysis — Primary comparisons are based on the MMRM LS Mean Value at week 12; Least Squares Mean Difference = -8.40

8. Secondary Outcome: Change From Baseline in Beta-Cell Function Using the Updated Homeostasis Model Assessment Beta-Cell Function (HOMA2-B) at 12 Weeks
Description: HOMA2-B is an estimated steady state beta cell function based on updated HOMA2 model. The HOMA2 model estimates steady state pancreatic beta cell function (%B) as a percentage of a normal reference population using simultaneously measured fasting plasma glucose and fasting insulin. Changes in HOMA2-B were analyzed by a mixed model repeated measures (MMRM) model that included dose, pre-study therapy, body mass index (BMI) group at baseline, baseline value, visit, and dose*visit, where the participant was treated as a random effect.
Time Frame: Baseline, 12 weeks
Population: Full analysis set: All randomized participants who received at least 1 dose of the study drug.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage beta-cell function
Arm/Group | 0.75 mg LY2189265 | 0.5 mg LY2189265 | 0.25 mg LY2189265 | Placebo
Number analyzed (Participants) | 32 | 32 | 33 | 33
percentage beta-cell function | 38.63 [29.36 to 47.90] | 26.67 [17.74 to 35.61] | 20.04 [11.19 to 28.89] | 6.94 [-2.10 to 15.98]
Statistical Analysis 1: Comparison: 0.75 mg LY2189265 vs 0.5 mg LY2189265 vs 0.25 mg LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — This is the p-value for the linear trend test at week 12
Statistical Analysis 2: Comparison: 0.25 mg LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.036, Mixed Models Analysis — Primary comparisons are based on the MMRM Least Squares (LS) Mean Value at week 12; Least Squares Mean Difference = 13.10
Statistical Analysis 3: Comparison: 0.5 mg LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis — Primary comparisons are based on the MMRM LS Mean Value at week 12; Least Squares Mean Difference = 19.73
Statistical Analysis 4: Comparison: 0.75 mg LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Primary comparisons are based on the MMRM LS Mean Value at week 12; Least Squares Mean Difference = 31.68

9. Secondary Outcome: Steady-State Concentrations of LY2189265
Description: Evaluable pharmacokinetics (PK) concentrations from all sampling time-points were combined and utilized in a population approach to determine the population mean estimate and standard deviation at 12 weeks. The model predicted LY2189265 steady state concentrations in each dose level were calculated as estimated area under the curve (AUC)/dosing period of 168 hours. The models and model parameters were described by nonlinear, mixed-effects regression modeling (NONMEM) using the program NONMEM 7®.
Time Frame: 12 weeks
Population: Full analysis set: All randomized participants who received at least 1 dose of the study drug.
Measure: Median (90% Confidence Interval); unit: nanograms per milliliter (ng/mL)
Groups:
- LY 0.25 mg: Administered by subcutaneous (SC) injection, once weekly (QW) for 12 weeks.
- LY 0.50 mg; LY 0.75 mg: Administered by SC injection, QW for 12 weeks.
Arm/Group | LY 0.25 mg | LY 0.50 mg | LY 0.75 mg
Number analyzed (Participants) | 36 | 36 | 34
nanograms per milliliter (ng/mL) | 15.8 [10.4 to 27.0] | 28.8 [19.2 to 47.4] | 42.7 [24.3 to 70.0]

10. Secondary Outcome: Percentage of Participants With Self-Reported Hypoglycemic Episodes During the 12-week Treatment Period
Description: Assessed the percentage of participants who reported a hypoglycemic episode during the 12-week treatment period. Hypoglycemia was defined as a measured plasma glucose level of ≤70 milligrams per deciliter (mg/dL) or ≤3.9 millimoles per liter (mmol/L).
Time Frame: 12 weeks
Population: Full analysis set: All randomized participants who received at least 1 dose of the study drug.
Measure: Number; unit: percentage of participants
Arm/Group | 0.75 mg LY2189265 | 0.5 mg LY2189265 | 0.25 mg LY2189265 | Placebo
Number analyzed (Participants) | 35 | 37 | 36 | 37
percentage of participants | 5.7 | 2.7 | 0.0 | 0.0
Statistical Analysis 1: Comparison: 0.75 mg LY2189265 vs 0.5 mg LY2189265 vs 0.25 mg LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.073, Cochran-Armitage — This is the p-value from the Cochran-Armitage trend test (dose-effect)
Statistical Analysis 2: Comparison: 0.5 mg LY2189265 vs Placebo; Test type: Superiority or Other; p = 1.00, Fisher Exact
Statistical Analysis 3: Comparison: 0.75 mg LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.233, Fisher Exact

ADVERSE EVENTS:
Groups:
- Placebo: Administered by subcutaneous (SC) injection, once weekly (QW) for 12 weeks.
- 0.75 mg LY2189265: Administered by SC injection, QW for 12 weeks.
Arm/Group | Placebo | 0.25 mg LY2189265 | 0.5 mg LY2189265 | 0.75 mg LY2189265
Serious Adverse Events (participants affected / at risk) | 0/37 | 1/36 | 0/37 | 1/35
Other Adverse Events (participants affected / at risk) | 16/37 | 17/36 | 18/37 | 15/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=37) | 0.25 mg LY2189265 (N=36) | 0.5 mg LY2189265 (N=37) | 0.75 mg LY2189265 (N=35)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VIIth nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=37) | 0.25 mg LY2189265 (N=36) | 0.5 mg LY2189265 (N=37) | 0.75 mg LY2189265 (N=35)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingivitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 6 (10) | 2 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperplastic cholecystopathy (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 6 (8) | 3 (4) | 3 (5) | 3 (3)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Electrocardiogram abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Intercostal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dyshidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral coldness (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days